CLINICAL TRIAL: NCT00266019
Title: Weight Management in Nonalcoholic Steatohepatitis (NASH)
Brief Title: Weight Management in Nonalcoholic Steatohepatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DK67363 (completed)
Record Dates: First submitted 2005-12-14; First posted 2005-12-15 (Estimated); Last update posted 2010-01-13 (Estimated); Status verified 2010-01

CONDITIONS: Fatty Liver
Keywords: nonalcoholic steatohepatitis; nonalcoholic fatty liver disease; Fatty liver; Cirrhosis; Obesity; Weight Reduction; Weight Management
MeSH Terms: conditions — Fatty Liver; Non-alcoholic Fatty Liver Disease; Fibrosis; Obesity; Weight Loss | interventions — Diet; Exercise; Behavior Therapy

INTERVENTIONS:
Behavioral: Weight Management (diet, exercise, and behavior modification)

SUMMARY:
Nonalcoholic steatohepatitis (NASH) is one of the most common chronic liver diseases. The cause of NASH is not completely understood and currently there is no effective treatment for this disease. An effective approach to treatment is needed since without treatment this disease may progress to fibrosis and cirrhosis. Obesity is one of the most important risk factors for NASH and weight reduction is generally recommended as an initial step in its management. However, there are very limited data on the efficacy of weight reduction as a treatment for NASH. Data from uncontrolled trials using poorly defined primary outcome measures and patient populations and nonstandardized weight loss interventions suggest that modest weight loss may improve fatty liver disease. The objective of this project is to conduct a randomized controlled trial of weight reduction in the management of NASH using a combination of diet, exercise, and behavior modification.

DETAILED DESCRIPTION:
Nonalcoholic steatohepatitis (NASH) is one of the most common chronic liver diseases. The cause of NASH is not completely understood and currently there is no effective treatment for this disease. An effective approach to treatment is needed since without treatment this disease may progress to fibrosis and cirrhosis. Obesity is one of the most important risk factors for NASH and weight reduction is generally recommended as an initial step in its management. However, there has never been a randomized controlled trial evaluating the efficacy of weight reduction as a treatment for NASH. Data from uncontrolled trials using poorly defined primary outcome measures and patient populations and nonstandardized weight loss interventions suggest that modest weight loss may improve liver histology. The objective of this project is to conduct a pilot study in preparation for a randomized controlled trial of weight reduction in the management of NASH. In this study, 30 overweight or obese individuals with biopsy-proven NASH will be enrolled. Twenty patients will be randomized to receive 48 weeks of intensive weight management using a combination of diet, exercise and behavior modification with a goal of 7-10% weight reduction. This weight loss program is similar to programs used successfully in other overweight populations and to the intensive lifestyle program of the Diabetes Prevention Program and Look AHEAD. The other 10 patients will be randomized to a control group where they will receive standard medical care and general counseling on healthy eating and exercise. At the end of the 48-week study, patients will have a repeat liver biopsy that will be compared to their baseline biopsy. The pilot study will establish the feasibility of recruiting and retaining, producing sustained weight loss and performing repeat liver biopsies in this population. Based on the outcomes of this preliminary trial, this program will be further refined and readied for a larger-scale clinical trial.

ELIGIBILITY:
Inclusion Criteria:

1. Evidence of chronic steatohepatitis on liver biopsy.
2. Elevated alanine or aspartate aminotransferase values (ALT > 41 or AST > 34) within 3 months of enrollment
3. Absence of another form of liver disease
4. Body mass index between 25-50 kg/m2.
5. At least 18 years of age
6. Absence of significant alcohol consumption (more than one standard drink per day).
7. Able to walk 2 blocks or a quarter of a mile without stopping
8. Willing to complete a two-week run-in period with successful completion of self-monitoring records.

Exclusion Criteria:

1. < 18 years of age
2. Significant alcohol consumption (> 1 standard drink per day)
3. Contraindications to obtaining a liver biopsy
4. Unable to walk 2 blocks or a quarter of a mile without stopping
5. Currently pregnant or pregnant in the previous six months
6. Currently engaged in an active weight-loss program or taking weight-loss medication
7. Report conditions that, in the judgment of the investigators, render potential participants unlikely to follow the protocol for 12 months, including illness likely to be terminal within 2 years, plans to move, substance abuse, or other significant psychiatric problems

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2005-01; Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Liver histology score (NASH-Clinical Research Network [CRN] scoring system) at 48 weeks
Weight reduction at 48 weeks

SECONDARY OUTCOMES:
Insulin sensitivity at 48 weeks
Liver function test at 48 weeks
Inflammatory markers and adipokine levels at 48 weeks
Quality of life at 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kittichai Promrat, M.D., Principal Investigator — Rhode Island Hospital/Brown University
Locations (1):
- Rhode Island Hospital, Providence, Rhode Island, United States

REFERENCES:
- [Background] Knowler WC, Barrett-Connor E, Fowler SE, Hamman RF, Lachin JM, Walker EA, Nathan DM; Diabetes Prevention Program Research Group. Reduction in the incidence of type 2 diabetes with lifestyle intervention or metformin. N Engl J Med. 2002 Feb 7;346(6):393-403. doi: 10.1056/NEJMoa012512. PMID 11832527
- [Background] Ludwig J, Viggiano TR, McGill DB, Oh BJ. Nonalcoholic steatohepatitis: Mayo Clinic experiences with a hitherto unnamed disease. Mayo Clin Proc. 1980 Jul;55(7):434-8. PMID 7382552
- [Background] Bacon BR, Farahvash MJ, Janney CG, Neuschwander-Tetri BA. Nonalcoholic steatohepatitis: an expanded clinical entity. Gastroenterology. 1994 Oct;107(4):1103-9. doi: 10.1016/0016-5085(94)90235-6. PMID 7523217
- [Background] Kleiner DE, Brunt EM, Van Natta M, Behling C, Contos MJ, Cummings OW, Ferrell LD, Liu YC, Torbenson MS, Unalp-Arida A, Yeh M, McCullough AJ, Sanyal AJ; Nonalcoholic Steatohepatitis Clinical Research Network. Design and validation of a histological scoring system for nonalcoholic fatty liver disease. Hepatology. 2005 Jun;41(6):1313-21. doi: 10.1002/hep.20701. PMID 15915461
- [Background] Ueno T, Sugawara H, Sujaku K, Hashimoto O, Tsuji R, Tamaki S, Torimura T, Inuzuka S, Sata M, Tanikawa K. Therapeutic effects of restricted diet and exercise in obese patients with fatty liver. J Hepatol. 1997 Jul;27(1):103-7. doi: 10.1016/s0168-8278(97)80287-5. PMID 9252081